CLINICAL TRIAL: NCT06412393
Title: Evaluation of Eye Health Benefits of Black Tomato Extract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS1-23170
Record Dates: First submitted 2024-05-03; First posted 2024-05-14 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Eye; High Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo powder (Placebo Comparator): Dietary Supplement: Placebo powder
  Interventions: Dietary Supplement: Placebo powder
- Black tomato extract powder (Experimental): Dietary Supplement: Black tomato extract powder
  Interventions: Dietary Supplement: Black tomato extract powder

INTERVENTIONS:
Dietary Supplement: Black tomato extract powder — take 2 packets per day for 8 weeks
  Arms: Black tomato extract powder
Dietary Supplement: Placebo powder — take 2 packets per day for 8 weeks
  Arms: Placebo powder

SUMMARY:
Verification of the efficacy of black tomato extract for eye health.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 20 and capable of providing informed consent.
* Daily usage of 3C (computer, communication, and consumer electronics) for more than 6 hours (OSDI screening - those experiencing dryness and fatigue in the eyes).
* BMI between 22 and 35.
* High myopia population (-5.00 to -9.00D)

Exclusion Criteria:

* History of any eye surgery (e.g., strabismus surgery, refractive surgery).
* Presence of systemic diseases affecting the anterior surface of the eye.
* Long-term use of medications affecting the anterior surface of the eye.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 56 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure Measurement (IOP) | Change from Baseline at 8 weeks
  Measurement of Intraocular Pressure using a non-contact tonometer. Unit: mmHg
Grading of Retinal Vascular Diameter | Change from Baseline at 8 weeks
  Measurement of Grading of Retinal Vascular Diameter using a fundus camera.
Visual Contrast Sensitivity Function | Change from Baseline at 8 weeks
  Perform the Visual Contrast Sensitivity Test (Distance and near) under environmental illumination/dark/bright conditions.
Negative Fusional Vergence (NFV) | Change from Baseline at 8 weeks
  Measurement of Negative Fusional Vergence using a phoropter.
Positive Fusional Vergence (PFV) | Change from Baseline at 8 weeks
  Measurement of Positive Fusional Vergence using a phoropter.
Negative Relative Accommodation (NRA) | Change from Baseline at 8 weeks
  Measurement of Negative Relative Accommodation using a phoropter.
Positive Relative Accommodation (PRA) | Change from Baseline at 8 weeks
  Measurement of Positive Relative Accommodation using a phoropter.
Accommodative Facility | Change from Baseline at 8 weeks
  Measurement of Accommodative Facility using a Flipper lens ±2.00D.

SECONDARY OUTCOMES:
Questionnaire Survey - Ocular Surface Disease Index (OSDI) | Change from Baseline at 8 weeks
  The OSDI is assessed on a scale of 0 to 100, with higher scores representing greater disability.
The change of Endothelin-1 (ET-1) | Change from Baseline at 8 weeks
  Fasting venous blood will be sampled to measure concentrations of ET-1.
The change of Tumor necrosis factor-α (TNF-α) | Change from Baseline at 8 weeks
  Fasting venous blood will be sampled to measure concentrations of TNF-α.
Best-corrected visual acuity | Change from Baseline at 8 weeks
  Measurement of Best-corrected visual acuity (distance and near) using a logMAR chart.

CONTACTS AND LOCATIONS:
Overall Officials: Bo-Yie Chen boychen@csmu.edu.tw, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan